CLINICAL TRIAL: NCT01524393
Title: Estimation of the Risk of Pulmonary Embolism and Venous Thromboembolism in Pregnancy After in Vitro Fertilization.
Brief Title: Risk of Pulmonary and Venous Thromboembolism in Pregnancies After in Vitro Fertilization
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Professor Peter Henriksson, Professor, Danderyd Hospital
Other Study IDs: Dnr 2010/267-31/4
Record Dates: First submitted 2012-01-28; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Pulmonary Embolism; Venous Thromboembolism
Keywords: Assisted Reproductive Techniques; Pregnancy; Pulmonary Embolism; Venous Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IVF pregnancy

SUMMARY:
Occurrence of venous thromboembolism during in Vitro Fertilization (IVF) pregnancies has been reported in numerous case reports and in two small consecutive series. The incidence of venous thromboembolism (VTE) after IVF has been claimed to be comparable to the incidence of VTE during normal pregnancy. No information exists concerning pulmonary embolism (PE).

The aim is to estimate and compare the risk of both PE and VTE during the the different phases of pregnancy after IVF to that in age and period matched control women. The investigators will use the Swedish National Health Registers to estimate the risk.

DETAILED DESCRIPTION:
Background: Occurrence of venous thromboembolism (VTE) during IVF pregnancies has been reported in numerous case reports and in two small consecutive series. The incidence of VTE after IVF has been claimed to be comparable to the incidence of VTE during normal pregnancy. No information exists concerning pulmonary embolism (PE).

Aim: The aim is to estimate and compare the risk of both PE and VTE during the trimesters of pregnancy after IVF to that in age and period matched control women.

Design and methods: A cross-sectional study using linkage of Swedish population and health registers. The Swedish National Patient Register encompasses inpatients and outpatients. Inpatient data in Sweden is available nationwide since 1987. Outpatient diagnoses from hospitals started to be collected in 1997. Data in the Patient Register will be linked to the Swedish Medical Birth Register (MBR) at the National Board of Health and Welfare through the unique personal identity number assigned to all Swedish residents, Exposed women: Mothers who had given birth to a child as a result of IVF will be retrieved from the Swedish IVF Register at the National Board of Health and Welfare. The Swedish IVF Register is now a part of the Swedish Medical Birth Register (MBR) at the National Board of Health and Welfare and includes information on IVF pregnancies since 1982.

We will restrict the retrieval to mothers of a child born as from 1990 until 2008 and who had their first child born after assisted reproduction by IVF.

Unexposed women: Each IVF woman will be matched with 5 unexposed women from the MBR by calendar year of delivery and maternal age.

Information will be retrieved on country of birth, pre-pregnancy body mass index, family situation, cigarette smoking habits, number of older siblings, singleton/multiple births, and estimated length of gestation from the MBR register. Dates of the trimesters is calculated from the length of gestation. Women´s education is found in the Register of Education, Statistics Sweden, by linkage through the personal identity number.

Diagnoses of VTE including PE will be found by linkage to the Swedish Patient Register of the National Board of Health and Welfare. This register comprises date of admission and discharge, and main diagnosis with up to seven contributing diagnoses. Diagnoses are recorded according to the International Classification of Diagnoses (ICD), ninth version prior to 1996 and the tenth version from 1997. Codes used were 415B, 451B, 452, 453C-D, 453W, 453X, 673C, 671D-E, 671F in ICD9 and I260, I269, I801- 3, I808-9, I822-3, I828-9, O223, O225, O871, O873, O879, O882 in ICD10.

The study is approved by the Research Ethics Committee of Karolinska Institutet, Stockholm, Sweden (Dnr 2010/267-31/4).

ELIGIBILITY:
Inclusion Criteria:

Exposed women:

* All mothers who had given birth to a child as a result of IVF will be retrieved from the Swedish Medical Birth Register (MBR) at the National Board of Health and Welfare.

Unexposed women:

* Each IVF woman will be matched with up to 5 unexposed women from the MBR by calendar year of delivery ±2 years and maternal age ±1 year.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All mothers who had given birth to a child.
Sampling Method: Non-Probability Sample
Enrollment: 140458 (Actual)
Dates: Start 1990-01; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Ekbom, Professor, Study Chair — Clinical Epidemiology Unit, Department of Medicine, Karolinska Institutet, Stockholm, Sweden; Peter Henriksson, Professor, Principal Investigator — Division of Cardiovascular Medicine, Department of Clinical Sciences, Danderyd Hospital, Karolinska Institutet, Stockholm, Sweden; Outi Hovatta, Professor, Study Chair — Department of Clinical Science, Intervention and Technology, Karolinska Institutet, Stockholm, Sweden
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Chan WS, Dixon ME. The "ART" of thromboembolism: a review of assisted reproductive technology and thromboembolic complications. Thromb Res. 2008;121(6):713-26. doi: 10.1016/j.thromres.2007.05.023. Epub 2007 Jul 30. PMID 17659766
- [Background] Mara M, Koryntova D, Rezabek K, Kapral A, Drbohlav P, Jirsova S, Zivny J. [Thromboembolic complications in patients undergoing in vitro fertilization: retrospective clinical study]. Ceska Gynekol. 2004 Jul;69(4):312-6. Czech. PMID 15369253
- [Derived] Henriksson P, Westerlund E, Wallen H, Brandt L, Hovatta O, Ekbom A. Incidence of pulmonary and venous thromboembolism in pregnancies after in vitro fertilisation: cross sectional study. BMJ. 2013 Jan 15;346:e8632. doi: 10.1136/bmj.e8632. PMID 23321489